CLINICAL TRIAL: NCT01809743
Title: Comparison of Regadenoson (Rapiscan) and Central Intravenous Adenosine for Measurement of Fractional Flow Reserve
Brief Title: Regadenoson and Adenosine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lokien van Nunen (Other)
Responsible Party: Sponsor-Investigator, Lokien van Nunen, MD, Catharina Ziekenhuis Eindhoven
Organization: Catharina Ziekenhuis Eindhoven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL42049.060.12
Record Dates: First submitted 2012-12-18; First posted 2013-03-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Regadenoson; Adenosine; Maximal hyperemia; Fractional flow reserve; FFR
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regadenoson central - peripheral (Active Comparator): First bolus regadenoson administered central, second bolus administered peripheral
  Interventions: Drug: Regadenoson central - peripheral; Drug: Adenosine
- Regadenoson peripheral - central (Active Comparator): First bolus regadenoson administered peripheral, second bolus administered central
  Interventions: Drug: Regadenoson peripheral - central; Drug: Adenosine
- Regadenoson central - central (Active Comparator): First bolus regadenoson administered central, second bolus administered central
  Interventions: Drug: Regadenoson central -central; Drug: Adenosine
- Regadenoson peripheral - peripheral (Active Comparator): First bolus regadenoson administered peripheral, second bolus administered peripheral
  Interventions: Drug: Regadenoson peripheral - peripheral; Drug: Adenosine

INTERVENTIONS:
Drug: Regadenoson central -central — To test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the golden standard).
  Arms: Regadenoson central - central
Drug: Regadenoson peripheral - peripheral — To test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the golden standard).
  Arms: Regadenoson peripheral - peripheral
Drug: Regadenoson central - peripheral — To test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the golden standard).
  Arms: Regadenoson central - peripheral
Drug: Regadenoson peripheral - central — To test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the golden standard).
  Arms: Regadenoson peripheral - central
Drug: Adenosine — Fractional flow reserve is measured by inducing hyperaemia using central adenosine infusion.

SUMMARY:
The aim of the study is to test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the gold standard)and to investigate the time intervals of maximum hyperemia induced by centrally and peripherally administered Regadenoson.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Scheduled for invasive measurement of FFR for diagnostic and interventional purposes in proximal or mid segments of a coronary artery

Exclusion Criteria:

* Severe aortic valve stenosis
* History of severe COPD
* Syncope or bradycardia (less than 50 beats/min)
* Known conduction disturbances (2nd-3rd degree heart-block, sick sinus without pacemaker or long QT-syndrome)
* Severe hypotension (RR <90 mmHg)
* Patients in whom no access to the coronary circulation can be obtained by the femoral artery or in whom femoral access was problematic
* Coronary anatomy not suitable for FFR measurement (extremely tortuous or calcified coronary vessels)
* Previous coronary bypass surgery
* Recent ST elevation myocardial infarction (<5 days)
* Recent non-ST elevation myocardial infarction (<5 days) if the peak CK is >1000 IU
* Inability to provide informed consent
* Pregnancy
* Use of methylxanthines (in the last 12 hours)
* Use of Dipyridamol (in the last 48 hours)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the accuracy of Regadenoson to induce maximal and steady state hyperemia | participants will be followed up during hospital stay, an expected average of 1 day
  To test the accuracy of Regadenoson to induce maximal and steady state hyperemia as compared to central venous infusion of adenosine for assessing fractional flow reserve. (adenosine is considered to be the gold standard).

SECONDARY OUTCOMES:
time intervals of maximum hyperemia | participants will be followed up during hospital stay, an expected average of 1 day
  To investigate the time intervals of maximum hyperemia induced by centrally and peripherally administered Regadenoson.

CONTACTS AND LOCATIONS:
Overall Officials: Nico H.J. Pijls, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; Lokien X van Nunen, MD, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

REFERENCES:
- [Derived] van Nunen LX, Lenders GD, Schampaert S, van 't Veer M, Wijnbergen I, Brueren GR, Tonino PA, Pijls NH. Single bolus intravenous regadenoson injection versus central venous infusion of adenosine for maximum coronary hyperaemia in fractional flow reserve measurement. EuroIntervention. 2015 Dec;11(8):905-13. doi: 10.4244/EIJY14M08_10. PMID 25136887